CLINICAL TRIAL: NCT01718769
Title: Validation of the STAMP Screening Tool For Pediatric Nutritional Risk To Be Used in the Ambulatory Setting.
Brief Title: Validation of the STAMP Screening Tool For Pediatric Nutritional Risk
Acronym: STAMP2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MMC206-2011KCTIL
Record Dates: First submitted 2012-03-20; First posted 2012-10-31 (Estimated); Last update posted 2016-04-27 (Estimated); Status verified 2015-04

CONDITIONS: Malnutrition
Keywords: Nutritional assessment; children; malnutrition
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- STAMP using (Active Comparator): 100 boys and girls aged 1 to 6, attending Clalit Health Care Services Pediatric Centers, will undergo an assessment using the STAMP Tool; a questionnaire including 3 questions with a summary score, according to which the nutritional risk level shall be determined. These children shall also undergo a complete dietician assessment in order to examine the validity of the STAMP Tool.
  Interventions: Other: questionnaire STAMP
- No STAMP using (Placebo Comparator): 150 files shall be reviewed in the beginning of the research and after 6 months in order to estimate the change in medical staff's attention to nutritional status, by way of noting relevant diagnoses, reference to nutritional status- related tests and recording of anthropometric measurements.
  Interventions: Other: questionnaire STAMP

INTERVENTIONS:
Other: questionnaire STAMP — Children will undergo an assessment using the STAMP Tool; a questionnaire including 3 questions with a summary score, according to which the nutritional risk level shall be determined. These children shall also undergo a complete dietician assessment in order to examine the validity of the STAMP Tool.

SUMMARY:
Background: Insufficient nutritional intake, with or without concomitant morbidity, leads to weight loss or insufficient weight gain, is related to an increase in morbidity and mortality and exposes the child to medical complications. In addition, obesity is also related to complications during hospitalization and complications in general, and therefore early identification of these children is extremely important. Studies show that malnutrition is frequent among children upon hospitalization, where the risk of pediatric nutritional deterioration increases, even in the presence of mild stress factors. This risk is frequent mainly among children that arrive at the hospital with an initial poor nutritional status. Improving the nutritional status as part of the standard of care already at the ambulatory setting might improve the prognosis of children when ill. In Israel, nutritional screening in not conducted among children since there is no proper validated screening tool. Study objectives: To test the accuracy of the STAMP Screening Tool for pediatric nutritional risk which is designed to be used by nurses, and to compare it to a complete nutritional assessment conducted by a dietician in Clalit Health Care Services clinics. In addition, the investigators wish to examine the effects of using a screening tool for nutritional risk on the medical staff's attention to the nutritional status; this is measured by the collection of nutritional status-related data and their recording in the patient file.

Methods: 100 boys and girls aged 1 to 6, attending Clalit Health Care Services Pediatric Centers, will undergo an assessment using the STAMP Tool; a questionnaire including 3 questions with a summary score, according to which the nutritional risk level shall be determined. These children shall also undergo a complete dietician assessment in order to examine the validity of the STAMP Tool. In addition, 150 files shall be reviewed in the beginning of the research and after 6 months in order to estimate the change in medical staff's attention to nutritional status, by way of noting relevant diagnoses, reference to nutritional status- related tests and recording of anthropometric measurements.

A statistical analysis to examine the validity of the STAMP Tool shall be carried out using the kappa test (K) (30). The effect of the STAMP Tool use shall be calculated using the chi square test.

ELIGIBILITY:
Inclusion Criteria:

1. children between 1 and 6 years old
2. children treated at the clinics participating in the study

Exclusion Criteria:

1. Lack of consent or lack of Hebrew proficiency
2. children that not receiving treatment in day hospitalization at any hospital

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2012-10; Primary Completion 2014-07 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Validity and reliability will be determined by comparing questionnaire scores with the complete nutritional assessment scores. | one year
  The STAMP questionnaire scores will be compared to a complete nutritional assessment conducted by a dietitian in Clalit Health Care Service clinics.
A change in frequency of recording of nutritional diagnoses for malnutrition; abnormal growth curves, FTT (Failure To Thrive), underweight, overweight, and obesity. | Baseline and after 1 year
  The following will be evaluated before and after conducting the study: % of children < percentile 5, % of children > percentile 85, % of children > percentile 95, frequency of referrals to a dietician, frequency of blood counts, frequency of tests: hemoglobin, transferrin and TLC, frequency of anemia, differences in infection diagnosis (pneumonia, UTI, etc.), frequency of referrals to the ER.

SECONDARY OUTCOMES:
To evaluate the frequency of malnutrition among children in the community in the study clinics. | one year
  The following will be measured: Height, weight and BMI recording,% of children > percentile 95 in the weight-height curve, frequency of referrals to a dietician, frequency of blood counts, frequency of tests: albumin, hemoglobin, transferrin and TLC, frequency of anemia, differences in infection diagnosis (pneumonia, UTI, etc.), frequency of referrals to the ER, exposure to professional material on the subject of nutrition (leaflets, videos) before and after intervention, change in the number of children under growth follow up by a multi-professional team.
To evaluate the ratio of children with acute or chronic malnutrition out of all malnourished children | one year
  The following will be measured: Height, weight and BMI recording,% of children > percentile 95 in the weight-height curve, frequency of referrals to a dietician, frequency of blood counts, frequency of tests: albumin, hemoglobin, transferrin and TLC, frequency of anemia, differences in infection diagnosis (pneumonia, UTI, etc.), frequency of referrals to the ER, exposure to professional material on the subject of nutrition (leaflets, videos) before and after intervention, change in the number of children under growth follow up by a multi-professional team.

CONTACTS AND LOCATIONS:
Overall Officials: Raanan Shamir, Professor, Principal Investigator — Institute of Gastroenterology, Nutrition and Liver Diseases, Schneider Children's Medical Center of Israel
Locations (1):
- Netka child healthcare services, Tel Aviv, Israel

REFERENCES:
- [Derived] Rub G, Marderfeld L, Poraz I, Hartman C, Amsel S, Rosenbaum I, Pergamentzev-Karpol S, Monsonego-Ornan E, Shamir R. Validation of a Nutritional Screening Tool for Ambulatory Use in Pediatrics. J Pediatr Gastroenterol Nutr. 2016 May;62(5):771-5. doi: 10.1097/MPG.0000000000001046. PMID 26628448